CLINICAL TRIAL: NCT02599194
Title: An Exploratory Study of the Role of 18F-FSPG PET/CT Imaging for Cancer Patients Receiving Therapy
Brief Title: 18F-FSPG PET/CT for Cancer Patients on Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrei Iagaru (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-31855; NCI-2015-01125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VARIMG0006 (Other: OnCore ID); P30CA124435 (NIH)
Record Dates: First submitted 2015-11-01; First posted 2015-11-06 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: B-Cell Neoplasm; Estrogen Receptor Negative; HER2/Neu Negative; Metastatic Renal Cell Cancer; Progesterone Receptor Negative; Stage III Mesothelioma; Stage III Renal Cell Cancer; Stage IIIA Breast Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Mesothelioma; Stage IV Non-Small Cell Lung Cancer; Stage IV Renal Cell Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Lymphoma, B-Cell; Carcinoma, Renal Cell; Mesothelioma; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — 4-(3-fluoropropyl)glutamic acid; (4S)-4-(3-(18F)fluoropropyl)-L-glutamate; Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Intra-patient comparison of 2 different radiolabels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FSPG and 18F-FDG Intragroup Comparision (Experimental): Participants sequentially receive radioimaging agents 18F-FSPG and 18F-FDG IV followed by PET/CT scan with 60 minutes.
  Interventions: Drug: 18F-FSPG; Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FSPG — Administered intravenously (IV)
  Other Names: 18F-labeled (S)-4-(3-[18F]-fluoropropyl)-L-glutamic acid; 18F-labeled (4S)-4-(3-[18F]-fluoropropyl)-L-glutamate; BAY94-9392
Drug: 18F-FDG — Administered intravenously (IV)
  Other Names: [18F]-Fluorodeoxyglucose ([18F]-FDG)

SUMMARY:
The goal of this phase 2 study trial is to evaluate the utility of the radiolabel 18F-FSPG used before and after treatment to diagnose, predict, and evaluate response to therapy in patients with a wide variety of metastatic cancers.

DETAILED DESCRIPTION:
OUTLINE:

Patients are evaluated with a PET/CT scan using the radiolabel 18F-FSPG [18F-(S)-4-(3-fluoropropyl)-L-glutamic acid] or 18F-FDG ([18F]-fluorodeoxyglucose), before and after therapeutic treatment.

PRIMARY OBJECTIVE:

Uptake of the radiolabel 18F-FSPG in patients with biopsy-proven cancer will be evaluated and compared to the uptake of 18F-FDG, before and after therapy (non-specified) in the same group of patients.

SECONDARY OBJECTIVES:

* Compare the agreement of the clinical assessment for cancer status between 18F-FSPG and 18F-FDG.
* Safety and tolerability of 18F-FSPG and 18F-FDG.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Able to complete a PET/CT scan without the use of sedation
* Females:

  * Of childbearing potential must:

    * Not be nursing
    * Have a negative serum pregnancy test documented within 48 hours prior to administration of 18F FSPG PET/CT
  * Not of childbearing potential must be:

    * Physiologically postmenopausal (cessation of menses for more than 1 year)
    * Surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy)
* Histologically confirmed cancer that is advanced; metastatic; or otherwise not suitable for surgical resection with curative intent
* Scheduled to begin therapy
* The time interval between 18F FSPG PET/CT and standard of care imaging (ie, 18F FDG PET/CT, diagnostic CT, or MRI) should be within 4 weeks (exceptions will be allowed for 6 weeks, if there are no other options)
* Ideally, there should be no chemotherapy, radiotherapy, or immune/biologic therapy or biopsy between other imaging (PET/CTs, MRI, or diagnostic CTs) and 18F FSPG PET/CT scheduled or performed (exceptions by investigator discretion)
* No clinically relevant deviations in renal function (serum creatinine > grade 2 Common Terminology Criteria for Adverse Events [CTCAE] version 4.0); maximal interval between confirmation of renal function and injection of 18F FSPG is 1 week

Exclusion Criteria:

* Scheduled for surgery and/or another invasive procedure (except biopsy) within the time period of 1 month prior to 18F FSPG administration
* Known sensitivity to 18F FSPG or components of the preparation
* Investigator precludes participation for scientific reasons, for reasons of compliance, or for reasons of the patient's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei M Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park P, Hatami N, Rutledge O, Koglin N, Loo B, Fan A, Mittra E. J Nucl Med. 58(suppl 1, no 118), 1 May 2017.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18F-FSPG and 18F-FDG Intragroup Comparision
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-FSPG and 18F-FDG Intragroup Comparision
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 69.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Standard Uptake Value Maximum (SUVmax) Post-treatment
Description: Standard Uptake Values (SUVs) for the radiotracers labels 18F-FSPG and 18F-FDG were assessed in tumor tissues of study participants, before (baseline), and after therapeutic treatment. Time frame was specified by protocol as at baseline, and at the time of clinical assessments during individual patient regular medical care. The time of the post-treatment assessment was not otherwise explicitly defined but could be anytime within 2 years. The outcome is reported as the difference of means from baseline to post-treatment (a number without dispersion), for all lesions for which an SUVmax value was assessed. A negative result indicates less uptake of radiotracer suggesting a small volume of tumor.
Time Frame: Baseline and up to 2 years
Population: Locations (ie, of lesions) that did not produce an SUVmax value either before or after treatment are omitted from the mean. Note that an analysis "mean of differences" would have a dispersion, but an analysis for "difference of means" is simply the delta (a number) between 2 measures of central tendency (mean), and does not have a dispersion.
Measure: Number; unit: g/mL
Units Other Than Participants: Lesion locations assessed
Arm/Group | 18F-FSPG and 18F-FDG Intragroup Comparision
Number analyzed (Participants) | 7
Number analyzed (Lesion locations assessed) | 40
g/mL
  18F-FSPG | -1.69
  18F-FDG | -0.64

2. Secondary Outcome: Number of Treatment-Related Adverse Events
Description: Safety and tolerability of 18F-FSPG and 18F-FDG were assessed as treatment-related adverse events, and reported as the number of events related to each treatment, without dispersion.
Time Frame: Baseline to up to 2 years
Measure: Number; unit: adverse events
Arm/Group | 18F-FSPG and 18F-FDG Intragroup Comparision
Number analyzed (Participants) | 7
adverse events
  18F-FSPG | 0
  18F-FDG | 0

3. Secondary Outcome: Change From Baseline in Lesion Size Post-treatment, by 18F-FSPG or 18F-FDGs
Description: Lesion size in centimeters (cm) were assessed in 2 dimensions from the computed tomography (CT) component of PET/CT and the area in cm2 calculated for lesion locations at baseline and after treatment. Time frame was specified by protocol as at baseline, and at the time of clinical assessments during individual patient regular medical care. The time of the post-treatment assessment was not otherwise explicitly defined but could be anytime within 2 years. The outcome is reported the difference in area in cm² for each lesion (a number without dispersion).
Time Frame: Baseline and up to 2 years
Population: * Lesion locations not detected both before and after treatment are reported as N/A for 2-D area (in the effect that an assessment could be made with the other radiolabel).
  * Lesions detected at either before or after treatment only are reported as the difference from zero.
Measure: Number; unit: cm2
Units Other Than Participants: Lesion locations assessed
Groups:
- Difference in Lesion Size as Detected by 18F-FSPG: Participants sequentially receive radioimaging agent 18F-FSPG IV followed by PET/CT scan with 60 minutes.
  18F-FSPG: Administered intravenously (IV)
- Difference in Lesion Size as Detected by 18F-FDG: Participants sequentially receive radioimaging agent 18F-FDG IV followed by PET/CT scan with 60 minutes.
  18F-FDG: Administered intravenously (IV)
Arm/Group | Difference in Lesion Size as Detected by 18F-FSPG | Difference in Lesion Size as Detected by 18F-FDG
Number analyzed (Participants) | 7 | 7
Number analyzed (Lesion locations assessed) | 17 | 26
cm2
  Adrenal / adrenal mass, left | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | 11.3
  Adrenal / hepatic dome | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -2.0
  Adrenal / liver metastatis | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -1.3
  Adrenal / lung base metastatis, lower lobe right | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | 1.4
  Adrenal / lung metastatis, left | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -0.7
  Lung / infrascapular subcut | 0.2 | NA — Lesion location was not detected by 18F-FDG both before and after treatment, and no difference can be reported for 2-D area.
  Lung / abdominal wall, upper quadrant right | 7.6 | 6.9
  Lung / adajcent subcarinal lymph node | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | 3.0
  Lung / aortopulmonary window lymph node | -1.1 | -2.8
  Lung / hilar lymph node, left | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -2.3
  Lung / infraspinatus mm, right | 10.4 | 10.2
  Lung / lingula nodule | -1.7 | -2.7
  Lung / mass, upper lobe left | -8.1 | -6.4
  Lung / mass, lower lobe right | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -14.5
  Lung / nodule 1, lower lobe right | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -0.8
  Lung / nodule 2, upper lobe right | -1.7 | -1.5
  Lung / nodule, upper lobe right | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -0.4
  Lung / paraesophageal lymph node | 0.9 | NA — Lesion location was not detected by 18F-FDG both before and after treatment, and no difference can be reported for 2-D area.
  Lung / post-basal, lower lobe right | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -3.6
  Lung / subcarinal lymph node | 1.4 | 11.4
  Renal / adrenal mass, right | 3.1 | 7.1
  Renal / aortopulmonary window lymph node, left | 1.1 | -1.2
  Renal / gluteal subcutaneous nodule | 0.2 | 0.2
  Renal / interlobar | 2.4 | NA — Lesion location was not detected by 18F-FDG both before and after treatment, and no difference can be reported for 2-D area.
  Renal / kidney midpole, right | -1.2 | -1.4
  Renal / omental nodule | -0.2 | 1.2
  Renal / paratracheal lymph node, right | 0.6 | -2.0
  Renal / parotid, right | NA — Lesion location was not detected by 18F-FSPG both before and after treatment, and no difference can be reported for 2-D area. | -2.3
  Renal / retroperitoneal lymph node, left | 1.6 | 2.2

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 18F-FSPG and 18F-FDG Intragroup Comparision
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-FSPG and 18F-FDG Intragroup Comparision (N=7)
Elevated blood ammonia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No